CLINICAL TRIAL: NCT01325935
Title: Optimal Duration of DAPT Following Treatment With Endeavor (Zotarolimus-eluting Stent) in Real-world Japanese Patients: A Prospective Multicenter Registry (OPERA)
Brief Title: Optimal Duration of DAPT Following Treatment With Endeavor (Zotarolimus-eluting Stent) in Real-world Japanese Patients
Acronym: OPERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Associations for Establishment of Evidence in Interventions (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPERA 1.0 - AEEI
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Disease; Cardiovascular Disease; Arteriosclerosis; Arterial Occlusive Disease; Vascular Disease; Clopidogrel; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short-term DAPT group (Experimental): 1,200 patients to be newly registered: Undergo 3-month (+ 30 days) DAPT (aspirin and clopidogrel)
  Interventions: Drug: Clopidogrel
- Long-term DAPT group (No Intervention): 1,200 patients to be appropriated from E-Japan post-marketing surveillance who meet all inclusion criteria and do not fall under any exclusion criteria of the present clinical study: Undergo 12-month DAPT (aspirin and clopidogrel)

INTERVENTIONS:
Drug: Clopidogrel — DAPT using aspirin 81 mg/day (minimal dose) and clopidogrel 75 mg/day should be conducted for 3 months (+ 30 days) after stenting.
  Arms: Short-term DAPT group

SUMMARY:
A prospective multicenter registry in real-world Japanese patients undergoing DAPT for three months after stenting. To assess the long-term safety of Endeavor Zotarolimus-eluting stent through noninferiority in the primary endpoint between two different continuous regimen (three and twelve months) groups of DAPT after stenting with Endeavor Zotarolimus-eluting stent in real-world Japanese patients and to examine the optimal duration of DAPT after stenting with Endeavor Zotarolimus-eluting stent. The long-term DAPT group in the present clinical study (to be appropriated from the post-marketing surveillance of Endeavor) should consist of consecutive patients undergoing DAPT for twelve months after stenting, while the short-term DAPT group (to be newly registered in the present clinical study) should consist of patients who are instructed to undergo DAPT for three months after stenting.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical inclusion criteria

   * Patient over age 20 years.
   * Patient who is clinically indicated for PCI by stenting at least in one coronary lesion that is visually confirmed by coronary angiography.
   * Patient who has agreed to conditions after receiving an explanation about the contents of the present clinical study and who has signed the consent form approved by the ethical review board at each study site.
   * Patient who has agreed to undergo all clinical FUs listed in the present protocol.
2. Coronary angiographic inclusion criteria:

   * Patient who has a > 50% occlusion or stenosis that is visually confirmed by coronary angiography in a native coronary artery > 2.5 mm in diameter and in whom the relevant coronary artery has an anatomical structure that is eligible for PCI with Endeavor Zotarolimus-eluting stent.

Exclusion Criteria:

1. Clinical exclusion criteria

   * Patient over age 85 years.
   * Patient with ST elevation MI who requires primary or rescue PCI and whose performance status falls under any of the exclusion criteria.
   * Patient with cardiogenic shock.
   * Patient who underwent stent treatment with BMS in other lesions within 6 months prior to the conduct of index PCI of the target vessel.
   * Patient who has undergone some treatment with DES for coronary lesions.
   * Patient who is scheduled to undergo elective surgery within 12 months after index PCI.
   * Patient whose left ventricular ejection fraction (LVEF) is < 40%.
   * Patient with a hemorrhagic predisposition or a history of coagulation abnormality
   * Patient in whom the total number of deployed stents exceeds 4,regardless of the number of lesions and the number of affected branches.
   * Patient with a verified history of CVA before stenting.
   * Patient with a verified history of active peptic ulcer or upper gastrointestinal tract bleeding before Stenting.
   * Patient showing impaired renal function. (serum creatinine concentration: > 1.8 mg/dL)
   * Patient with known contraindications for aspirin or clopidogrel. (the physician should assess tolerability within the range of routine medical care)
   * Patient with a known disorder who has a life expectancy of less than 12 months.
   * Patient who is incompetent to adhere to all clinical FUs listed in the present protocol.
2. Angiographic exclusion criteria:

   * Lesions located within the saphenous venin graft (SVG).
   * Unprotected lesions in the left coronary trunk.
   * Lesions of in-stent restenosis in previously deployed DES or BMS.
   * Lesions with an anatomical structure of the coronary artery that is not eligible for treatment by the deployment of Endeavor ZES.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1187 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
NACCE (Net adverse clinical and cerebral event) | 12 months
  NACCE is defined as a composite endpoint consisting of death from some causes (including cardiac death and noncardiac death), myocardial infarction (Q-wave MI and non-Q wave MI), cerebral vascular accident, and major bleeding (as per the modified version of REPLACE-2 criteria for bleeding and as per GUSTO criteria for bleeding).

SECONDARY OUTCOMES:
Stent thrombosis | 12 months
  Incidence of stent thrombosis as per the definition by academic research council
MACE (major adverse cardiac events) | 1, 3, 6, 9 and 12 months
  Incidence of MACE at months 1, 3, 6, 9, and 12 after stenting. MACE is defined as a composite endpoint consisting of cardiac death from some causes (including cardiac and noncardiac death), MI (Q-wave MI and non-Q wave MI), TLR, and coronary artery bypass graft (CABG).
TVR (target vessel revascularization) | 9 and 12 months
  Incidence of target vessel revascularization at months 9 and 12 after stenting.
TLR (target lesion revascularization) | 9 and 12 months
  Incidence of target lesion revascularization at months 9 and 12 after stenting.
DAPT compliance | 12 months
  Duration of DAPT and patient compliance.
Hemorrhagic complications | 12 months
  Incidence of hemorrhagic complications. (as per the modified version of REPLACE-2 criteria for bleeding and as per GUSTO criteria for bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Takaaki Isshiki, M.D., Principal Investigator — Teikyo University; Shinsuke Nanto, M.D., Principal Investigator — Osaka University; Masato Nakamura, M.D., Principal Investigator — Toho University Ohashi Medical Center
Locations (112):
- Japan (112):
  - Asahi General Hospital, Asahi, Chiba
  - Kimitsu Chuo Hospital, Kisarazu, Chiba
  - Fukui Cardiovascular Center, Fukui-shi, Fukui
  - Fukuoka City Hospital, Fukuoka, Fukuoka
  - Fukuoka City Medical Association Hospital, Fukuoka, Fukuoka
  - Fukuoka Red Cross Hospital, Fukuoka, Fukuoka
  - University of Occupational and Environmental Health, Kita-Kyushu City, Fukuoka
  - National Hospital Organization Fukuoka-Higashi Medical Center, Koga, Fukuoka
  - Gifu Heart Center, Gifu, Gifu
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - Hiroshima Railway Hospital, Hiroshima, Hiroshima
  - Tsuchiya General Hospital, Hiroshima, Hiroshima
  - Engaru-Kosei General Hospital, Monbetsu-gun, Hokkaido
  - Hyogo Prefectural Amagasaki Hospital, Amagasaki, Hyōgo
  - Kansai Rosai Hospital, Cardiovascular Center, Amagasaki, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Shakaihoken Kobe Central Hospital, Kobe, Hyōgo
  - Miki City Hospital, Miki, Hyōgo
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Meiwa General Hospital, Nishinomiya, Hyōgo
  - Hyogo Prefectural Awaji Hospital, Sumoto, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kaisei General Hospital, Sakaidechō, Kagawa-ken
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Tenyoukai Central Hospital, Kagoshima, Kagoshima-ken
  - Ebina General Hospital, Ebina, Kanagawa
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Kawasaki Municipal Tama Hospital, Kawasaki, Kanagawa
  - St. Marianna University of Medicine, Toyoko Hospital, Kawasaki, Kanagawa
  - St. Marianna University School of Medicine, Kawasaki, Kanagawa
  - Synthesis Shinkawahashi Hospital, Kawasaki, Kanagawa
  - Odawara Cardiovascular Hospital, Odawara, Kanagawa
  - Kitazato University School of Medicine, Sagamihara, Kanagawa
  - Sagamihara Kyodo Hospital, Sagamihara, Kanagawa
  - Kanagawa Cardiovascular and Reppiratory Center, Yokohama, Kanagawa
  - Saiseikai Yokohama Tobu Hospital, Yokohama, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - St. Marianna University of Medicine, Yokohama City West Hospital, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Yokohama City UNiversity Medical Center, Yokohama, Kanagawa
  - Kumamoto Chuo Hospital, Kumamoto, Kumamoto
  - Kumamoto Red Cross Hospital, Kumamoto, Kumamoto
  - National Hospital Organization Kumamoto Medical Center, Kumamoto, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Sugimura Hospital, Kumamoto, Kumamoto
  - Ijinkai Takeda General Hospital, Kyoto, Kyoto
  - Koseikai Takeda Hospital, Kyoto, Kyoto
  - Kyoto Second Red Cross Hospital, Kyoto, Kyoto
  - Gakken The Holy City Medical Association Hospital, Sagara-gun, Kyoto
  - Uji Tokushukai Hospital, Uji, Kyoto
  - Matsuzaka Central General Hospital, Matsuzaka City, Mie-ken
  - Suzuka Central General Hospital, Suzuka, Mie-ken
  - Mie Heart Center, Taki-gun, Mie-ken
  - Mie University Hospital, Tsu, Mie-ken
  - Nagasaki University Graduate School of Biomedical Science, Nagasaki, Nagasaki
  - Kawasaki Medical School, Kurashiki, Okayama-ken
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - The Sakakibara Heart Institute of Okayama, Okayama, Okayama-ken
  - Ohama Daiichi Hospital, Naha, Okinawa
  - Nakagami Hospital, Okinawa, Okinawa
  - Okinawa Nanbu Tokushukai Hospital, Shimajiri-gun, Okinawa
  - Urasoe General Hospital, Urasoe, Okinawa
  - Kawachi General Hospital, Higashiosaka, Osaka
  - Kansai Medical University Hirakata Hospital, Hirakata, Osaka
  - Kansai Medical University Takii Hospital, Moriguchi, Osaka
  - Komatsu General Hospital, Neyagawa, Osaka
  - Higashi-sumiyoshi Morimoto Hospital, Osaka, Osaka
  - Nissay Hospital, Osaka, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka City University, Graduate School of Medicine, Osaka, Osaka
  - Osaka Ekisaikai Hospital, Osaka, Osaka
  - Osaka General Hospital of West Japan Railway Campany, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka Gyoumeikan Hospital, Osaka, Osaka
  - Osaka Police Hospital, Osaka, Osaka
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Bell Land General Hospital, Sakai, Osaka
  - Mimihara General Hospital, Sakai, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Osaka University Graduate School of Medicine, Suita, Osaka
  - Saiseikai Senri Hospital, Suita, Osaka
  - Hokusetsu General Hospital, Takatsuki, Osaka
  - Midorigaoka Hospital, Takatsuki, Osaka
  - Department of Cardiovascular Medicine, Saga University, Saga, Saga-ken
  - Mashiko Hospital, Kawaguchi, Saitama
  - Saitama Medical Center, Jichi Medical University, Saitama, Saitama
  - Kusatsu Heart Center, Kusatsu, Shiga
  - Shiga Medical Center for Adults, Moriyama, Shiga
  - Omihachiman Community Medical Center, Ōmihachiman, Shiga
  - Biwako Ohashi Hospital, Ōtsu, Shiga
  - Hamamatsu Medical Center, Hamamatsu, Shizuoka
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Shizuoka Hospital, Izunokuni, Shizuoka
  - Tokushima Red Cross Hospital, Komatsushimachō, Tokushima
  - Ayase Heart Hospital, Adachi-ku, Tokyo
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Tokyo Metroporitan Tama Medical Center, Fuchū, Tokyo
  - Itabashi Chuo Medical Center, Itabashi-ku, Tokyo
  - Nihon University School of Medicine, Itabashi-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Tokyo Metroporitan Geriatric Hospital and Institute of Gerontology, Itabashi-ku, Tokyo
  - Toho University Medical Center Ohashi Hospital, Meguro-ku, Tokyo
  - The Cardiovascular Institute, Minato-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - JR Tokyo General Hospital, Shibuya-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Tottri University, Yonago, Tottri
  - Shuto General Hospital, Yanai, Yamaguchi
  - Non-profit organization Associations for Establishiment of Evidence in Interventions, Minato-ku, Tokyo